CLINICAL TRIAL: NCT05819073
Title: Astringency Perception and Oral Health
Brief Title: Astringency and Oral Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Beverly J Tepper, Ph.D., Professor, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro2022000271
Record Dates: First submitted 2022-10-28; First posted 2023-04-19 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Saliva Altered; Taste, Altered
MeSH Terms: conditions — Dysgeusia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROP non-taster subjects (Experimental): This arm will comprise of PROP non-taster subjects. Subjects will use a cranberry-derived oral rinse twice a day for 11 days following a 3-day plain water-rinse period.
  Interventions: Other: Plain water; Other: CPE
- PROP super-taster subjects (Experimental): This arm will comprise of PROP super-taster subjects. Subjects will use a cranberry-derived oral rinse twice a day for 11 days following a 3-day plain water-rinse period.
  Interventions: Other: Plain water; Other: CPE

INTERVENTIONS:
Other: Plain water — Subjects will use plain water as an oral rinse twice a day for 3 days.
Other: CPE — Subjects will use a cranberry-derived oral rinse twice a day for 11 days.

SUMMARY:
The perception of astringency is thought to involve the interaction between tannins and salivary proteins. However, the mechanisms underlying this interaction are poorly understood. The tannins' subclass known as type A proanthocyanidins seems to have a positive effect on human health. Despite that, humans show large individual differences in the sensory perception and acceptance of astringent foods such as tea, wine and chocolate suggesting that this variation may have a genetic basis. Salivary proteins play an essential role both in affecting oral taste perception and in maintaining a healthy oral environment. Diverse microorganisms inhabit the oral cavity. The interactions between oral microbiota, host and environmental factors influence microbial homeostasis and ultimately human oral health. Understanding individual differences in salivary proteins, oral microbiome and the mechanisms by which tannins evoke the perception of astringency could provide important insights into the role of these compounds in human nutrition and health.

DETAILED DESCRIPTION:
This study examines the effects of a daily Cranberry Polyphenol Extract (CPE) oral rinse on salivary protein responses and the oral microbiome (as a proxy measure of oral health). The study will be conducted in healthy adults who are presumably at high-risk or low-risk of oral disease. High risk individuals include non-tasters of PROP (6-n-propylthiouracil) and homozygous recessive for TAS2R38 (Taste 2 Receptor Member 38) gene, while low-risk individuals include super-tasters of PROP and homozygous dominant for TAS2R38 gene.

The specific aims are to determine if the use of cranberry polyphenol extract rinse will:

1. alter the oral microbial profile
2. induce changes in the salivary protein response
3. be associated with changes in taste and flavor perception

Participants will be screened for good overall and oral health. Each subject's period of participation will be 2 weeks. Days 1-3 of the study is a run-in period. Subjects will rinse with spring water 2-times/day (after brushing their teeth in the morning and evening). During days 4-14, subjects will rinse in a similar manner with a solution of CPE in spring water. Saliva will be collected from subjects in a brief session (10 min) on day 1, day 3, and day 14. Saliva samples will be analyzed for gene, salivary proteins and microbial profile analysis. The purpose of this analysis is to measure the relative ratios of beneficial vs. disease-causing microbes in the mouth using microbial whole-genome sequencing (WGS). On each of the testing days, subjects will also evaluate food samples for standard taste and flavor attributes.

ELIGIBILITY:
Inclusion Criteria:

* PROP insensitive individuals (PROP non-tasters; homozygous recessive for TAS2R38 gene)
* PROP high-sensitive individuals (PROP super-tasters; homozygous dominant for TAS2R38 gene)
* Overall healthy; good oral health and hygiene routine
* Current on a routine checkup by a oral/dental health professional
* Recently underwent dental/cleaning by a oral/dental health professional
* No ongoing oral health problems
* Agree to use intervention material as prescribed
* Agree to refrain from using any other oral rinse material during the term of the study

Exclusion Criteria:

* PROP medium-taster individuals (heterozygous for TAS2R38 gene)
* Taste or smell dysfunction
* Pregnant or nursing
* Oral piercings
* Smoking
* Use of medications other than birth control

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Taste and Flavor Intensity Ratings after 11 days | Baseline measure 3 days after control intervention; Post intervention measure 11 days after experimental intervention
  Taste and flavor intensity ratings of cranberry juice and aronia juice samples will be collected 3 days after control intervention and then at the end of the experimental intervention. An end-anchored (None, Very Strong) 15 cm line scale will be used with taste and key flavor attributes.
Change from Baseline Levels of Salivary Proteins after 11 days | Baseline measure 3 days after control intervention; Post intervention measure 11 days after experimental intervention
  Saliva will be collected 3 days after control intervention and then at the end of the experimental intervention. Samples will be analyzed via dot blot analysis and LC-MS (liquid chromatography-mass spectrometry) to establish proteomic composition before and after the intervention. Specifically, area of the ion current peaks (XIC peaks) generated will be used as a relative quantity of the salivary protein levels. The XIC peaks are proportional to the concentration of salivary proteins under constant conditions and will be used to understand the effect of the intervention on salivary protein levels.
Change from Baseline Composition of Oral Microbiome after 11 days | Baseline measure 3 days after control intervention; Post intervention measure 11 days after experimental intervention
  Salivary samples will be collected 3 days after control intervention and then at the end of the experimental intervention. Samples will be analyzed for microbial composition via Whole Genome Sequencing and data used to understand changes in microbial diversity before and after the intervention. Specifically operational taxonomic units will be identified and classified at the species level.

CONTACTS AND LOCATIONS:
Overall Officials: Beverly J Tepper, Ph.D., Principal Investigator — Rutgers University
Locations (1):
- Rutgers University, Department of Food Science, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after de-identification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning three months and ending 5 years after publication.
Access Criteria: Anyone who wishes to access the data. For any purpose.

DOCUMENTS (1):
  • Informed Consent Form (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT05819073/ICF_000.pdf